CLINICAL TRIAL: NCT00159393
Title: Percutaneous Nephrolithotomy: A Registry and Database
Status: Completed | Type: Observational
Sponsor: Indiana Kidney Stone Institute (Other)
Responsible Party: Principal Investigator, James Lingeman, Director, Indiana Kidney Stone Institute
Other Study IDs: 03-096
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Nephrolithiasis
Keywords: Kidney stones; nephrolithotripsy percutaneous
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: registry and database — data collection

SUMMARY:
Kidney stones vary in size from a tiny grain of sand to as large as filling the inside of the kidney. Treatment decisions depend on the size, location, and composition of the stone. Some kidney stones can be treated with lithotripsy (breaking up stones inside the body with shock waves created outside the body) or ureteroscopy (placing a small telescope up the urine channel to remove the stone). When stones are large in size or in the lower part of the kidney, a percutaneous (making a passage from the back into the kidney) procedure has been found to be the best method to remove the stones safely and efficiently. A passage is made into the back to allow a small telescope to see the stone and break it into fragments for removal. A small catheter is placed at the end of the procedure to allow the kidney to drain.

The purpose of this study is to record information about your surgery into a database so we can look at how patients who have had this procedure have done over time. We hope that reporting the outcomes of this surgery will be helpful to urologists and patients in the future. There may be certain factors that can be identified through this study as having better outcomes that may help make future surgeries safer.

DETAILED DESCRIPTION:
Patients of IU Health Physicians Urology who have been scheduled to undergo percutaneous removal of one or more kidney stones will be asked to consent to be part of our registry and database for percutaneous procedures. The database contains information about the subjects surgery, such as stone size and location, number of access sites to remove the stone, length of stay in the hospital, secondary procedures, etc. This information is reviewed periodically to look for trends so that physicians may find ways to improve the percutaneous procedure. All information in the database is kept confidential. Data is collected at follow-up appointments at one month and one year to see if the subject is still stone free.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients of Methodist Urology in Indianapolis, IN
* Male or female patients with upper urinary tract stone disease appropriate for percutaneous removal as determined by a Methodist Urology physician

EXCLUSION CRITERIA:

* Patients unable to give informed consent
* Patients with active bleeding diatheses
* Women who are pregnant or in whom pregnancy status cannot be confirmed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: urology clinic patients already scheduled for percutaneous removal of kidney stones
Sampling Method: Non-Probability Sample
Enrollment: 1697 (Actual)
Dates: Start 2003-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — IU Health Physicians Urology
Locations (2):
- United States (2):
  - Indiana University Health, Carmel, Indiana
  - IU Health North Hospital, Carmel, Indiana

REFERENCES:
- [Background] Kim SC, Kuo RL, Lingeman JE. Percutaneous nephrolithotomy: an update. Curr Opin Urol. 2003 May;13(3):235-41. doi: 10.1097/00042307-200305000-00012. PMID 12692448